CLINICAL TRIAL: NCT01341314
Title: Proof of Concept of an Internet-based Series Design Case-finding System for Very Early Rheumatoid Arthritis.
Brief Title: Finding Early Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Matthew H. Liang, MD, Principal Investigator, Brigham and Women's Hospital
Other Study IDs: ArthFndtn
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Joint Pain; Stiffness
Keywords: joint pain; stiffness
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen serum for future assay development
Oversight: Data Monitoring Committee: No

SUMMARY:
Research has shown that early aggressive use of medicines may stop rheumatoid arthritis (RA)or slow its damage. The key to this is to find people with early symptoms which could be RA and have them get a diagnosis, treatment and follow-up.

This study will recruit persons who've gone to the internet looking for information about their symptoms. After answering a screening survey, the person with possible symptoms will be linked to the study website for a more detailed symptom questionnaire.

After completing that questionnaire the person will receive information about the second part of the study which includes an examination with a rheumatologist (arthritis doctor)and laboratory tests.

Based on the joint examination and laboratory tests, the rheumatologist will tell the person the likelihood of having RA, and make recommendations and if needed a referral for care and treatment. Treatment is not a part of this study.

This study will also compare the information on the subject's questionnaires to the doctor's joint examination and the laboratory tests with the hope of developing a simple inexpensive case finding questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Joint pain or swelling for less than 3 months
* Be able to use the internet

Exclusion Criteria:

* Non English speaking
* Diagnosis of rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: persons with joint pain or swelling for less than 3 months
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2010-01; Primary Completion 2013-01 (Estimated); Study Completion 2013-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States